CLINICAL TRIAL: NCT04097275
Title: Induced Pluripotent Stem Cells for the Development of Novel Drug Therapies for Inborn Errors of Metabolism, an International, Multicenter Study
Brief Title: Induced Pluripotent Stem Cells for the Development of Novel Drug Therapies for Inborn Errors of Metabolism (iPSC-IEM)
Acronym: iPSC-IEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: iPSC-IEM-2019
Record Dates: First submitted 2019-08-23; First posted 2019-09-20 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Inborn Errors of Metabolism
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with an Inborn Error of Metabolism
  Interventions: Other: Skin biopsy; Other: Withdraw of blood

INTERVENTIONS:
Other: Skin biopsy — The biopsy will be performed by means of punch biopsy (diameter 2.5 mm) under local anesthesia on a forearm. The skin biopsy will be transferred to sterile cell culture Dulbecco's Modified Eagle Medium (DMEM) 1% Penicillin 1% Streptomycin 1% Gentamycin medium 10% FBS.
Other: Withdraw of blood — Blood will be collected in:
  * 1 x Ethylene Diamine Tetraacetic Acid (EDTA) tube (7.5 ml) - for further leucocytes extraction that are a potential backup for new iPS cell lines generation
  * 1 x Citrate Phosphate Dextrose Adenine (CPDA) tube (8.5 ml) - for EBV-transformed lymphoblastoid cell lines generation
  * 1 x Dried Blood Spot DBS-filtercard, called CentoCard® - for quality control confirmatory genetic testing

SUMMARY:
Human induced pluripotent stem cells (iPSCs), are reprogrammed from somatic cells that can self-renew indefinitely and produce different types of cells. They provide human model cell lines for orphan drug development. It is the goal of this study to define new cellular disease models for Inborn Erors of Metabolism, as enabling tools for both drug discovery and development.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant or from the parent/ legal guardian
* The participant is aged between 2 months and 50 years
* The diagnosis of an Inborn Error of Metabolism (IEM) is genetically confirmed by Centogene
* The participant is a first-degree or a second-degree relative of an individual with Inborn Error of Metabolism (IEM) genetically confirmed by Centogene

Exclusion Criteria:

* Inability to provide informed consent
* The participant is younger than 2 months or older than 50 years
* The diagnosis of an Inborn Error of Metabolism (IEM) is not genetically confirmed by Centogene and
* The participant is not a first-degree or a seconddegree relative of an individual with Inborn Error of Metabolism (IEM) genetically confirmed by Centogene
* Previously enrolled in the study

Ages: 2 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with an Inborn Error of Metabolism
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Generation of patient-specific induced pluripotent stem cells and then differentiate them into neural cells. | 1 day
  To generate patient-specific induced pluripotent stem cells and then differentiate them into neural cells, or other specific cell according to the Inborn Error of Metabolism, to study the misfolded proteins in endoplasmic reticulum, their role in untranslated protein response, and possible mechanisms to shuttle the misfolded proteins into lysosomes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (1):
- Children Hospital and Institute of Child Health, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No